CLINICAL TRIAL: NCT02980692
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose, Phase 2b Study to Demonstrate the Safety and Efficacy of Tildrakizumab in Subjects With Active Psoriatic Arthritis
Brief Title: Efficacy and Safety Study of SUNPG1623
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLR_16_23
Record Dates: First submitted 2016-11-30; First posted 2016-12-02 (Estimated); Results first posted 2021-05-19 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2022-08

CONDITIONS: Active Psoriatic Arthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- SUNPG1623 dose I (Experimental): low range dose
  Interventions: Drug: SUNPG1623 I
- SUNPG1623 dose II (Experimental): mid range dose
  Interventions: Drug: SUNPG1623 II; Drug: PLACEBO
- SUNPG1623 dose III (Experimental): mid range dose
  Interventions: Drug: SUNPG1623 III; Drug: PLACEBO
- SUNPG1623 dose IV (Experimental): mid range dose to high dose
  Interventions: Drug: SUNPG1623 IV; Drug: PLACEBO
- Placebo (Placebo Comparator): mid range dose to high dose
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: SUNPG1623 I — injection
  Arms: SUNPG1623 dose I
Drug: SUNPG1623 II — injection
  Arms: SUNPG1623 dose II
Drug: SUNPG1623 III — injection
  Arms: SUNPG1623 dose III
Drug: SUNPG1623 IV — injection
  Arms: SUNPG1623 dose IV
Drug: PLACEBO — injection
  Arms: Placebo; SUNPG1623 dose II; SUNPG1623 dose III; SUNPG1623 dose IV

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multiple-dose, phase 2b study to demonstrate the safety and efficacy of SUNPG1623

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided written informed consent
* Subject is ≥ 18 years of age at time of Screening
* Subject must be on stable dose of NSAID for ≥ 4 weeks prior to initiation of IMP
* Subject has a negative evaluation for TB within 4 weeks before initiating IMP
* Subject has a diagnosis of PsA (by the Classification of Psoriatic Arthritis [CASPAR] criteria) with symptoms present for at least 6 months.
* Subject has ≥ 3 tender and ≥ 3 swollen joints at Screening and Baseline.

Exclusion Criteria:

* Subject has a planned surgical intervention between Baseline and the Week 24 evaluation for a pretreatment condition
* Subject has an active infection or history of infections
* Subject has any concurrent medical condition or uncontrolled, clinically significant systemic disease
* Subject has a known history of infection with hepatitis B, hepatitis C, or human immunodeficiency virus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 391 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-09-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- SPARC Site 1, Middleburg Heights, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mease PJ, Chohan S, Fructuoso FJG, Luggen ME, Rahman P, Raychaudhuri SP, Chou RC, Mendelsohn AM, Rozzo SJ, Gottlieb A. Efficacy and safety of tildrakizumab in patients with active psoriatic arthritis: results of a randomised, double-blind, placebo-controlled, multiple-dose, 52-week phase IIb study. Ann Rheum Dis. 2021 Sep;80(9):1147-1157. doi: 10.1136/annrheumdis-2020-219014. Epub 2021 May 13. PMID 33985942

RESULTS

PARTICIPANT FLOW:
Groups:
- SUNPG1623 I: Group: SUNPG1623 I dosage: Short-term dose dosage form: subcutaneous injection frequency of administration: q4 weeks
- SUNPG1623 II: Group: SUNPG1623 II dosage: Mid-term dose dosage form: subcutaneous injection frequency of administration: q12 weeks
- SUNPG1623 Dose III: Group: SUNPG1623 III dosage: Mid-term dose dosage form: subcutaneous injection frequency of administration: q12 weeks
- SUNPG1623 Dose IV: Group: SUNPG1623 IV dosage: Mid to long-term dose dosage form: subcutaneous injection frequency of administration: q12 weeks
  Subjects who received SUNPG1623 Dose IV during Part 1 but failed to show clinical response to treatment at Week 24 entered Part 2 and received SUNPG1623 II until Week 48
- Placebo: Group: Placebo dosage: Mid to long-term dose dosage form: subcutaneous injection frequency of administration: q12 weeks
  Subjects who received placebo during Part 1 but failed to show clinical response to treatment at Week 24 entered Part 2 and received SUNPG1623 II until Week 48
Period: Double Blind Placebo Controlled Period
Arm/Group | SUNPG1623 I | SUNPG1623 II | SUNPG1623 Dose III | SUNPG1623 Dose IV | Placebo
Started | 78 | 79 | 77 | 78 | 79
Completed | 62 | 64 | 60 | 71 | 74
Not Completed | 16 | 15 | 17 | 7 | 5
Not completed — Adverse Event | 1 | 2 | 1 | 2 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 1 | 0
Not completed — Investigator Decision | 0 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 2 | 4
Not completed — Protocol Violation | 2 | 0 | 1 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 0 | 1
Not completed — Failure to show sufficient response to treatment at Week 24 | 9 | 12 | 13 | 0 | 0
Period: Double-blind Follow-up Period
Arm/Group | SUNPG1623 I | SUNPG1623 II | SUNPG1623 Dose III | SUNPG1623 Dose IV | Placebo
Started | 62 | 64 | 60 | 71 | 74
Completed | 62 | 61 | 56 | 67 | 69
Not Completed | 0 | 3 | 4 | 4 | 5
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1
Not completed — Failure to show sufficient response to treatment at Week 24 | 0 | 2 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 1
Not completed — Other | 0 | 0 | 1 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SUNPG1623 I | SUNPG1623 II | SUNPG1623 Dose III | SUNPG1623 Dose IV | Placebo | Total
Number analyzed (Participants) | 78 | 79 | 77 | 78 | 79 | 391
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (13.28) | 49.3 (11.24) | 49.2 (11.85) | 47.2 (13.35) | 48.1 (13.30) | 48.8 (12.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 37 | 47 | 41 | 44 | 215
  Male | 32 | 42 | 30 | 37 | 35 | 176
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 16 | 11 | 9 | 11 | 59
  Not Hispanic or Latino | 66 | 63 | 66 | 69 | 68 | 332
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1 | 3 | 5
  White | 76 | 78 | 75 | 75 | 74 | 378
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 1 | 2 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Who Achieve American College of Rheumatology20 Response Rate
Description: The American College of Rheumatology20 response measured the percentage of subjects with at least a 20% improvement from Baseline in both tender joints (68) and swollen joints (66) and a 20% improvement in three of the following five criteria: patient global assessment, physician global assessment, patient pain assessment, patient self-assessed disability, and acute-phase C-reactive protein.
  For 'Units of Measure'- Data entered is proportion of participants, which is calculated by dividing the value obtained (percentage in this case) by 100.
Time Frame: week 24
Population: Cochran-Mantel-Haenszel Analysis of ACR20 Response Rate At Week 24 (Missing Response = Non-response) - Primary Analysis (Full Analysis Set)
Measure: Number; unit: proportion of subjects
Groups:
- SUNPG1623 Dose IV: Group: SUNPG1623 IV dosage: Mid to long-term dose dosage form: subcutaneous injection frequency of administration: q12 weeks
- Placebo: Group: Placebo dosage: Mid to long-term dose dosage form: subcutaneous injection frequency of administration: q12 weeks
Arm/Group | SUNPG1623 I | SUNPG1623 II | SUNPG1623 Dose III | SUNPG1623 Dose IV | Placebo
Number analyzed (Participants) | 78 | 79 | 77 | 78 | 79
proportion of subjects | 0.7949 | 0.7722 | 0.7143 | 0.7308 | 0.5063
Statistical Analysis 1: Comparison: SUNPG1623 I vs Placebo; Test type: Superiority; p = 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: SUNPG1623 II vs Placebo; Test type: Superiority; p = 0.0006, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: SUNPG1623 Dose III vs Placebo; Test type: Superiority; p = 0.0088, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: SUNPG1623 Dose IV vs Placebo; Test type: Superiority; p = 0.0041, Cochran-Mantel-Haenszel

2. Secondary Outcome: Proportion of Subjects Who Achieve American College of Rheumatology20 Response Rate
Description: as for outcome 1
Time Frame: week 52
Population: Full Analysis Set
Measure: Number; unit: proportion of subjects
Groups:
- SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24: Group: SUNPG1623 IV dosage: Mid to long-term dose dosage form: subcutaneous injection frequency of administration: q12 weeks
  Subjects who received SUNPG1623 Dose IV during Part 1 but failed to show clinical response to treatment at Week 24 entered Part 2 and received SUNPG1623 II until Week 48
- Placebo Moved to SUNPG1623 II After Week 24: Group: Placebo dosage: Mid to long-term dose dosage form: subcutaneous injection frequency of administration: q12 weeks
  Subjects who received placebo during Part 1 but failed to show clinical response to treatment at Week 24 entered Part 2 and received SUNPG1623 II until Week 48
Arm/Group | SUNPG1623 I | SUNPG1623 II | SUNPG1623 Dose III | SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24 | Placebo Moved to SUNPG1623 II After Week 24
Number analyzed (Participants) | 67 | 64 | 60 | 75 | 75
proportion of subjects | 0.9254 | 0.8906 | 0.8667 | 0.8133 | 0.8133
Statistical Analysis 1: Comparison: SUNPG1623 I; Test type: Superiority; % response rate = 92.54, 95% CI 2-sided [86.24 to 98.83], Standard Error of Mean 3.21
Statistical Analysis 2: Comparison: SUNPG1623 II; Test type: Superiority; % response rate = 89.06, 95% CI 2-sided [81.42 to 96.71], Standard Error of Mean 3.90
Statistical Analysis 3: Comparison: SUNPG1623 Dose III; Test type: Superiority; % response rate = 86.67, 95% CI 2-sided [78.07 to 95.27], Standard Error of Mean 4.39
Statistical Analysis 4: Comparison: SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24; Test type: Superiority; % response rate = 81.33, 95% CI 2-sided [72.52 to 90.15], Standard Error of Mean 4.50
Statistical Analysis 5: Comparison: Placebo Moved to SUNPG1623 II After Week 24; Test type: Superiority; % response rate = 81.33, 95% CI 2-sided [72.52 to 90.15], Standard Error of Mean 4.50

3. Secondary Outcome: Proportion of Subjects Achieving American College of Rheumatology50 Response Rate
Description: The American College of Rheumatology50 response measured the percentage of subjects with at least a 50% improvement from Baseline in both tender joints (68) and swollen joints (66) and a 50% improvement in three of the following five criteria: patient global assessment, physician global assessment, patient pain assessment, patient self-assessed disability, and acute-phase C-reactive protein.
  For 'Units of Measure'- Data entered is proportion of participants, which is calculated by dividing the value obtained (percentage in this case) by 100.
Time Frame: week 1, week 4, week 8, week 12, week 16, week 20, week 24 and week 52
Population: Cochran-Mantel-Haenszel Analysis of ACR50 Response Rates up to Week 24 Full Analysis Set.
  ACR50 Response Rates up to Week 52 Full Analysis Set.
Measure: Number; unit: proportion of subjects
Arm/Group | SUNPG1623 I | SUNPG1623 II | SUNPG1623 Dose III | SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24 | Placebo Moved to SUNPG1623 II After Week 24
Number analyzed (Participants) | 78 | 79 | 77 | 78 | 79
proportion of subjects
  Week 1 | 0 | 0.0253 | 0.0130 | 0.0128 | 0
  Week 4 | 0.0256 | 0.0506 | 0.0909 | 0.0385 | 0.0253
  Week 8 | 0.1667 | 0.0759 | 0.1299 | 0.1410 | 0.0759
  Week 12 | 0.1795 | 0.1772 | 0.2078 | 0.1923 | 0.0633
  Week 16 | 0.3077 | 0.2785 | 0.2727 | 0.2051 | 0.0506
  Week 20 | 0.4487 | 0.4177 | 0.2857 | 0.2308 | 0.1646
  Week 24 | 0.5256 | 0.5063 | 0.4545 | 0.3974 | 0.2405
  week 52: number analyzed (Participants) | 67 | 64 | 61 | 75 | 75
  week 52 | 0.7910 | 0.7500 | 0.7213 | 0.6800 | 0.6267
Statistical Analysis 1: Comparison: SUNPG1623 I; Test type: Superiority; % response rate = 79.10, 95% CI 2-sided [69.37 to 88.84], Standard Error of Mean 4.97
Statistical Analysis 2: Comparison: SUNPG1623 II; Test type: Superiority; % response rate = 75.00, 95% CI 2-sided [64.39 to 85.61], Standard Error of Mean 5.41
Statistical Analysis 3: Comparison: SUNPG1623 Dose III; Test type: Superiority; % response rate = 72.13, 95% CI 2-sided [60.88 to 83.38], Standard Error of Mean 5.74
Statistical Analysis 4: Comparison: SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24; Test type: Superiority; % response rate = 68.00, 95% CI 2-sided [57.44 to 78.56], Standard Error of Mean 5.39
Statistical Analysis 5: Comparison: Placebo Moved to SUNPG1623 II After Week 24; Test type: Superiority; % response rate = 62.67, 95% CI 2-sided [51.72 to 73.61], Standard Error of Mean 5.59

4. Secondary Outcome: Proportion of Subjects Achieving American College of Rheumatology70 Response Rate
Description: The American College of Rheumatology70 response measured the percentage of subjects with at least a 50% improvement from Baseline in both tender joints (68) and swollen joints (66) and a 50% improvement in three of the following five criteria: patient global assessment, physician global assessment, patient pain assessment, patient self-assessed disability, and acute-phase C-reactive protein.
  For 'Units of Measure'- Data entered is proportion of participants, which is calculated by dividing the value obtained (percentage in this case) by 100.
Time Frame: week 1, week 4, week 8, week 12, week 16, week 20, week 24, and week 52
Population: Cochran-Mantel-Haenszel Analysis of ACR70 Response Rates up to Week 24 Full Analysis Set ACR70 Response Rates up to Week 52 Full Analysis Set.
Measure: Number; unit: proportion of subjects
Arm/Group | SUNPG1623 I | SUNPG1623 II | SUNPG1623 Dose III | SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24 | Placebo Moved to SUNPG1623 II After Week 24
Number analyzed (Participants) | 78 | 79 | 77 | 78 | 79
proportion of subjects
  Week 1 | 0 | 0.0127 | 0 | 0 | 0
  Week 4 | 0.0128 | 0.0127 | 0 | 0.0128 | 0.0127
  Week 8 | 0.0256 | 0.0380 | 0.0260 | 0.0256 | 0.0380
  Week 12 | 0.1026 | 0.0380 | 0.0649 | 0.1026 | 0.0127
  Week 16 | 0.1410 | 0.1266 | 0.1169 | 0.0897 | 0.0253
  Week 20 | 0.2051 | 0.2658 | 0.1429 | 0.1282 | 0.0380
  Week 24 | 0.2821 | 0.2911 | 0.2208 | 0.1667 | 0.1013
  week 52: number analyzed (Participants) | 67 | 64 | 61 | 75 | 75
  week 52 | 0.5821 | 0.4844 | 0.3934 | 0.4000 | 0.3733
Statistical Analysis 1: Comparison: SUNPG1623 I; Test type: Superiority; % response rate = 58.21, 95% CI 2-sided [46.40 to 70.02], Standard Error of Mean 6.03
Statistical Analysis 2: Comparison: SUNPG1623 II; Test type: Superiority; % response rate = 48.44, 95% CI 2-sided [36.19 to 60.68], Standard Error of Mean 6.25
Statistical Analysis 3: Comparison: SUNPG1623 Dose III; Test type: Superiority; % response rate = 39.34, 95% CI 2-sided [27.09 to 51.60], Standard Error of Mean 6.25
Statistical Analysis 4: Comparison: SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24; Test type: Superiority; % response rate = 40.00, 95% CI 2-sided [28.91 to 51.09], Standard Error of Mean 5.66
Statistical Analysis 5: Comparison: Placebo Moved to SUNPG1623 II After Week 24; Test type: Superiority; % response rate = 37.33, 95% CI 2-sided [26.39 to 48.28], Standard Error of Mean 5.59

5. Secondary Outcome: Change From Baseline in Tender Joint Counts
Description: Peripheral joints were assessed for tenderness and swelling. There is no validated measure to assess peripheral joints in Psoriatic arthritis; the measure used was the American College of Rheumatology joint count initially developed for the assessment of patients with rheumatoid arthritis.
Time Frame: week 1, week 4, week 8, week 12, week 16, week 20, and week 24
Measure: Least Squares Mean (Standard Error); unit: tender joint counts
Arm/Group | SUNPG1623 I | SUNPG1623 II | SUNPG1623 Dose III | SUNPG1623 Dose IV | Placebo
Number analyzed (Participants) | 77 | 78 | 76 | 78 | 79
tender joint counts
  Week 1 | -1.5 (0.77) | -2.4 (0.76) | -2.5 (0.78) | -3.1 (0.76) | -2.1 (0.76)
  Week 4 | -4.7 (0.89) | -4.9 (0.88) | -5.4 (0.89) | -3.9 (0.88) | -4.1 (0.87)
  Week 8 | -7.1 (0.94) | -7.8 (0.92) | -8.6 (0.94) | -7.2 (0.93) | -6.9 (0.91)
  Week 12 | -8.3 (0.96) | -10.0 (0.94) | -8.7 (0.95) | -7.8 (0.96) | -7.7 (0.94)
  Week 16 | -10.3 (1.04) | -11.3 (1.01) | -10.7 (1.03) | -9.8 (1.04) | -8.4 (1.02)
  Week 20 | -11.2 (1.09) | -12.3 (1.06) | -11.5 (1.07) | -11.4 (1.09) | -9.9 (1.06)
  Week 24 | -11.9 (1.04) | -12.6 (1.01) | -12.9 (1.03) | -12.0 (1.04) | -9.4 (1.02)
Statistical Analysis 1: Comparison: SUNPG1623 I vs Placebo; Test type: Superiority; p = 0.0850, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: SUNPG1623 II vs Placebo; Test type: Superiority; p = 0.0234, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: SUNPG1623 Dose III vs Placebo; Test type: Superiority; p = 0.0140, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: SUNPG1623 Dose IV vs Placebo; Test type: Superiority; p = 0.0731, Cochran-Mantel-Haenszel

6. Secondary Outcome: Change From Baseline in Tender Joint Counts
Description: as for outcome 5
Time Frame: Week 52
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: tender joint counts
Arm/Group | SUNPG1623 I | SUNPG1623 II | SUNPG1623 Dose III | SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24 | Placebo Moved to SUNPG1623 II After Week 24
Number analyzed (Participants) | 78 | 79 | 77 | 78 | 79
tender joint counts | -12.3 (11.47) | -13.7 (11.92) | -16.0 (12.83) | -14.0 (10.65) | -13.9 (12.02)
Statistical Analysis 1: Comparison: SUNPG1623 I; Test type: Superiority; Mean Difference (Net) = -12.3, Standard Deviation 11.47
Statistical Analysis 2: Comparison: SUNPG1623 II; Test type: Superiority; Mean Difference (Net) = -13.7, Standard Deviation 11.92
Statistical Analysis 3: Comparison: SUNPG1623 Dose III; Test type: Superiority; Mean Difference (Net) = -16.0, Standard Deviation 12.83
Statistical Analysis 4: Comparison: SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24; Test type: Superiority; Mean Difference (Net) = -14.0, Standard Deviation 10.65
Statistical Analysis 5: Comparison: Placebo Moved to SUNPG1623 II After Week 24; Test type: Superiority; Mean Difference (Net) = -13.9, Standard Deviation 12.02

7. Secondary Outcome: Change From Baseline in Swollen Joint Counts
Description: as for outcome 5
Time Frame: week 1, week 4, week 8, week 12, week 16, week 20, and week 24
Population: Statistical Analysis (Mixed Model Repeated Measures) of Change From Baseline in Swollen Joint Counts up to Week 24 - (No Imputation) Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Swollen Joint Counts
Arm/Group | SUNPG1623 I | SUNPG1623 II | SUNPG1623 Dose III | SUNPG1623 Dose IV | Placebo
Number analyzed (Participants) | 77 | 78 | 76 | 78 | 79
Swollen Joint Counts
  Week 1 | -1.8 (0.51) | -2.1 (0.51) | -1.3 (0.52) | -2.4 (0.51) | -1.3 (0.51)
  Week 4 | -4.1 (0.56) | -3.8 (0.55) | -3.8 (0.56) | -3.0 (0.55) | -3.1 (0.55)
  Week 8 | -5.8 (0.55) | -5.5 (0.54) | -5.7 (0.55) | -5.0 (0.55) | -4.7 (0.54)
  Week 12 | -7.3 (0.55) | -6.6 (0.54) | -6.2 (0.55) | -4.8 (0.55) | -4.9 (0.54)
  Week 16 | -8.0 (0.56) | -7.2 (0.55) | -7.0 (0.55) | -6.0 (0.56) | -5.2 (0.55)
  Week 20 | -8.3 (0.56) | -7.4 (0.55) | -7.4 (0.56) | -6.8 (0.56) | -6.0 (0.55)
  Week 24 | -8.3 (0.52) | -7.7 (0.51) | -8.2 (0.52) | -7.6 (0.52) | -6.5 (0.51)
Statistical Analysis 1: Comparison: SUNPG1623 I vs Placebo; Test type: Superiority; p = 0.0111, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: SUNPG1623 II vs Placebo; Test type: Superiority; p = 0.0774, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: SUNPG1623 Dose III vs Placebo; Test type: Superiority; p = 0.0190, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: SUNPG1623 Dose IV vs Placebo; Test type: Superiority; p = 0.1282, Cochran-Mantel-Haenszel

8. Secondary Outcome: Change From Baseline in Swollen Joint Counts
Description: as for outcome 5
Time Frame: Week 52
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Swollen Joint Counts
Arm/Group | SUNPG1623 I | SUNPG1623 II | SUNPG1623 Dose III | SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24 | Placebo Moved to SUNPG1623 II After Week 24
Number analyzed (Participants) | 78 | 79 | 77 | 78 | 79
Swollen Joint Counts | -8.7 (6.88) | -7.5 (7.07) | -9.2 (7.62) | -7.5 (5.78) | -9.0 (8.80)
Statistical Analysis 1: Comparison: SUNPG1623 I; Test type: Superiority; Mean Difference (Net) = -8.7, Standard Deviation 6.88
Statistical Analysis 2: Comparison: SUNPG1623 II; Test type: Superiority; Mean Difference (Net) = -7.5, Standard Deviation 7.07
Statistical Analysis 3: Comparison: SUNPG1623 Dose III; Test type: Superiority; Mean Difference (Net) = -9.2, Standard Deviation 7.62
Statistical Analysis 4: Comparison: SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24; Test type: Superiority; Mean Difference (Net) = -7.5, Standard Deviation 5.78
Statistical Analysis 5: Comparison: Placebo Moved to SUNPG1623 II After Week 24; Test type: Superiority; Mean Difference (Net) = -9.0, Standard Deviation 8.80

9. Secondary Outcome: Physician Global Assessment of Disease Activity Visual Analog Scale
Description: 100 mm Visual analog scale with descriptors (verbal) : "very good" (0) to "very poor" (100)
Time Frame: week 1, week 4, week 8, week 12, week 16, week 20, and week 24
Measure: Least Squares Mean (Standard Error); unit: scores on a visual analog scale
Arm/Group | SUNPG1623 I | SUNPG1623 II | SUNPG1623 Dose III | SUNPG1623 Dose IV | Placebo
Number analyzed (Participants) | 77 | 78 | 76 | 78 | 79
scores on a visual analog scale
  Week 1 | -7.8 (1.69) | -8.0 (1.68) | -7.2 (1.70) | -6.2 (1.68) | -4.5 (1.67)
  Week 4 | -14.3 (2.01) | -15.7 (1.99) | -15.1 (1.99) | -14.0 (1.99) | -9.7 (1.95)
  Week 8 | -21.9 (2.20) | -23.6 (2.16) | -23.9 (2.18) | -20.8 (2.18) | -16.2 (2.13)
  Week 12 | -27.9 (2.22) | -28.7 (2.17) | -27.6 (2.19) | -23.1 (2.22) | -18.5 (2.17)
  Week 16 | -31.0 (2.08) | -32.1 (2.03) | -31.7 (2.05) | -30.8 (2.08) | -20.2 (2.04)
  Week 20 | -36.7 (2.19) | -36.8 (2.13) | -31.0 (2.15) | -33.0 (2.19) | -24.3 (2.13)
  Week 24 | -36.5 (2.15) | -38.8 (2.08) | -37.5 (2.11) | -36.3 (2.14) | -23.5 (2.09)
Statistical Analysis 1: Comparison: SUNPG1623 I vs Placebo; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: SUNPG1623 II vs Placebo; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: SUNPG1623 Dose III vs Placebo; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: SUNPG1623 Dose IV vs Placebo; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel

10. Secondary Outcome: Change From Baseline in Physician Global Assessment of Disease Activity Visual Analog Scale
Description: 100 mm Visual analog scale with descriptors (verbal) : "very good" (0) to "very poor" (100)
Time Frame: Week 52
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: scores on a visual analog scale
Arm/Group | SUNPG1623 I | SUNPG1623 II | SUNPG1623 Dose III | SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24 | Placebo Moved to SUNPG1623 II After Week 24
Number analyzed (Participants) | 78 | 79 | 77 | 78 | 79
scores on a visual analog scale | -40.0 (17.38) | -44.3 (19.73) | -45.3 (19.84) | -42.7 (19.18) | -42.0 (20.41)
Statistical Analysis 1: Comparison: SUNPG1623 I; Test type: Superiority; Mean Difference (Net) = -40.0, Standard Deviation 17.38
Statistical Analysis 2: Comparison: SUNPG1623 II; Test type: Superiority; Mean Difference (Net) = -44.3, Standard Deviation 19.73
Statistical Analysis 3: Comparison: SUNPG1623 Dose III; Test type: Superiority; Mean Difference (Net) = -45.3, Standard Deviation 19.84
Statistical Analysis 4: Comparison: SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24; Test type: Superiority; Mean Difference (Net) = -42.7, Standard Deviation 19.18
Statistical Analysis 5: Comparison: Placebo Moved to SUNPG1623 II After Week 24; Test type: Superiority; Mean Difference (Net) = -42.0, Standard Deviation 20.41

11. Secondary Outcome: Patient's Global Assessment of Disease Activity
Description: 100 mm Visual analog scale descriptors (verbal) : "very well" (0) to "very poorly"(100)
Time Frame: week 1, week 4, week 8, week 12, week 16, week 20 and week 24
Measure: Least Squares Mean (Standard Error); unit: scores on a visual analog scale
Arm/Group | SUNPG1623 I | SUNPG1623 II | SUNPG1623 Dose III | SUNPG1623 Dose IV | Placebo
Number analyzed (Participants) | 77 | 78 | 76 | 78 | 79
scores on a visual analog scale
  Week 1 | -5.9 (1.85) | -7.5 (1.84) | -6.8 (1.87) | -6.4 (1.84) | -2.8 (1.84)
  Week 4 | -7.5 (2.17) | -11.9 (2.14) | -9.5 (2.15) | -8.8 (2.14) | -5.9 (2.11)
  Week 8 | -15.4 (2.30) | -15.5 (2.25) | -14.5 (2.28) | -13.1 (2.28) | -10.1 (2.23)
  Week 12 | -18.1 (2.52) | -20.3 (2.46) | -16.1 (2.49) | -16.4 (2.51) | -11.2 (2.46)
  Week 16 | -23.5 (2.63) | -22.0 (2.57) | -18.7 (2.59) | -19.4 (2.63) | -13.8 (2.58)
  Week 20 | -29.7 (2.64) | -27.3 (2.57) | -22.7 (2.60) | -21.6 (2.64) | -15.6 (2.58)
  Week 24 | -35.0 (2.60) | -33.3 (2.52) | -33.4 (2.56) | -30.4 (2.60) | -21.7 (2.54)
Statistical Analysis 1: Comparison: SUNPG1623 I vs Placebo; Test type: Superiority; p = 0.0003, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: SUNPG1623 II vs Placebo; Test type: Superiority; p = 0.0012, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: SUNPG1623 Dose III vs Placebo; Test type: Superiority; p = 0.0011, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: SUNPG1623 Dose IV vs Placebo; Test type: Superiority; p = 0.0167, Cochran-Mantel-Haenszel

12. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Disease Activity
Description: 100 mm Visual analog scale descriptors (verbal) : "very well" (0) to "very poorly"(100)
Time Frame: Week 52
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: scores on a visual analog scale
Arm/Group | SUNPG1623 I | SUNPG1623 II | SUNPG1623 Dose III | SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24 | Placebo Moved to SUNPG1623 II After Week 24
Number analyzed (Participants) | 78 | 79 | 77 | 78 | 79
scores on a visual analog scale | -42.2 (22.74) | -43.8 (24.01) | -38.4 (27.90) | -37.9 (24.65) | -40.5 (28.13)
Statistical Analysis 1: Comparison: SUNPG1623 I; Test type: Superiority; Mean Difference (Net) = -42.2, Standard Deviation 22.74
Statistical Analysis 2: Comparison: SUNPG1623 II; Test type: Superiority; Mean Difference (Net) = -43.8, Standard Deviation 24.01
Statistical Analysis 3: Comparison: SUNPG1623 Dose III; Test type: Superiority; Mean Difference (Net) = -38.4, Standard Deviation 27.90
Statistical Analysis 4: Comparison: SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24; Test type: Superiority; Mean Difference (Net) = -37.9, Standard Deviation 24.65
Statistical Analysis 5: Comparison: Placebo Moved to SUNPG1623 II After Week 24; Test type: Superiority; Mean Difference (Net) = -40.5, Standard Deviation 28.13

13. Secondary Outcome: Patient's Pain Assessment
Description: 100 mm Visual Analog Scale with scale (verbal descriptors) "no pain" (0) to "worst possible pain" (100).
Time Frame: week 1, week 4, week 8, week 12, week 16, week 20, and week 24
Population: Statistical Analysis (Mixed Model Repeated Measures) of Change From Baseline in Patient's Pain Assessment up to Week 24 - (No Imputation) Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: scores on a visual analog scale
Arm/Group | SUNPG1623 I | SUNPG1623 II | SUNPG1623 Dose III | SUNPG1623 Dose IV | Placebo
Number analyzed (Participants) | 77 | 78 | 76 | 78 | 79
scores on a visual analog scale
  Week 1 | -5.8 (1.96) | -8.1 (1.95) | -5.1 (1.98) | -5.8 (1.95) | -1.6 (1.95)
  Week 4 | -9.8 (2.15) | -12.8 (2.12) | -8.9 (2.13) | -6.4 (2.12) | -3.9 (2.09)
  Week 8 | -16.9 (2.42) | -16.1 (2.37) | -16.6 (2.41) | -11.9 (2.40) | -8.5 (2.35)
  Week 12 | -19.4 (2.54) | -20.4 (2.48) | -15.6 (2.50) | -14.0 (2.53) | -11.5 (2.48)
  Week 16 | -23.8 (2.58) | -23.2 (2.52) | -20.6 (2.55) | -19.3 (2.59) | -12.8 (2.54)
  Week 20 | -29.8 (2.79) | -25.3 (2.71) | -21.4 (2.74) | -21.4 (2.78) | -17.1 (2.72)
  Week 24 | -35.1 (2.69) | -31.6 (2.60) | -32.1 (2.64) | -28.8 (2.68) | -21.5 (2.63)
Statistical Analysis 1: Comparison: SUNPG1623 I vs Placebo; Test type: Superiority; p = 0.0003, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: SUNPG1623 II vs Placebo; Test type: Superiority; p = 0.0055, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: SUNPG1623 Dose III vs Placebo; Test type: Superiority; p = 0.0039, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: SUNPG1623 Dose IV vs Placebo; Test type: Superiority; p = 0.0487, Cochran-Mantel-Haenszel

14. Secondary Outcome: Change From Baseline in Patient's Pain Assessment
Description: 100 mm Visual Analog Scale with scale (verbal descriptors) "no pain" (0) to "worst possible pain" (100).
Time Frame: Week 52
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: scores on a visual analog scale
Arm/Group | SUNPG1623 I | SUNPG1623 II | SUNPG1623 Dose III | SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24 | Placebo Moved to SUNPG1623 II After Week 24
Number analyzed (Participants) | 78 | 79 | 77 | 78 | 79
scores on a visual analog scale | -40.7 (21.59) | -42.7 (25.67) | -38.0 (29.26) | -37.6 (26.63) | -41.0 (29.83)
Statistical Analysis 1: Comparison: SUNPG1623 I; Test type: Superiority; Mean Difference (Net) = -40.7, Standard Deviation 21.59
Statistical Analysis 2: Comparison: SUNPG1623 II; Test type: Superiority; Mean Difference (Net) = -42.7, Standard Deviation 25.67
Statistical Analysis 3: Comparison: SUNPG1623 Dose III; Test type: Superiority; Mean Difference (Net) = -38.0, Standard Deviation 29.26
Statistical Analysis 4: Comparison: SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24; Test type: Superiority; Mean Difference (Net) = -37.6, Standard Deviation 26.63
Statistical Analysis 5: Comparison: Placebo Moved to SUNPG1623 II After Week 24; Test type: Superiority; Mean Difference (Net) = -41.0, Standard Deviation 29.83

15. Secondary Outcome: Health Assessment Questionnaire- Disability Index
Description: eight categories assessed by the Health Assessment Questionnaire - Disability Index 1) dressing and grooming, 2) arising, 3) eating, 4) walking, 5) hygiene, 6) reach, 7) grip and 8) common daily activities was scored as 0 (without any difficulty), 1 (with some difficulty), 2 (with much difficulty) or 3 (unable to do).
  The score for the disability index is the mean of the 8 category scores. If more than 2 of the categories, or 25%, are missing, the scale is not scored. If fewer than 2 of the categories are missing, the sum of the categories is divided by the number of answered categories. A higher score indicates greater disability
Time Frame: week 1, week 4, week 8, week 12, week 16, week 20, and week 24
Measure: Least Squares Mean (Standard Error); unit: score for the disability index
Arm/Group | SUNPG1623 I | SUNPG1623 II | SUNPG1623 Dose III | SUNPG1623 Dose IV | Placebo
Number analyzed (Participants) | 77 | 78 | 76 | 78 | 79
score for the disability index
  Week 1 | -0.0374 (0.03454) | -0.0453 (0.03436) | -0.0552 (0.03492) | -0.0411 (0.03435) | -0.0045 (0.03439)
  Week 4 | -0.0025 (0.04036) | -0.0736 (0.03984) | -0.0906 (0.03999) | -0.0409 (0.03989) | -0.0404 (0.03928)
  Week 8 | -0.1510 (0.04709) | -0.1279 (0.04627) | -0.2035 (0.04687) | -0.1041 (0.04669) | -0.1265 (0.04588)
  Week 12 | -0.1310 (0.04601) | -0.2140 (0.04507) | -0.2090 (0.04555) | -0.1731 (0.04597) | -0.1374 (0.04503)
  Week 16 | -0.2061 (0.04890) | -0.2448 (0.04790) | -0.2343 (0.04843) | -0.2102 (0.04889) | -0.1580 (0.04801)
  Week 20 | -0.3052 (0.05256) | -0.2868 (0.05128) | -0.2911 (0.05185) | -0.1947 (0.05244) | -0.2271 (0.05135)
  Week 24 | -0.3013 (0.05196) | -0.3314 (0.05054) | -0.3337 (0.05128) | -0.2376 (0.05187) | -0.1827 (0.05102)
Statistical Analysis 1: Comparison: SUNPG1623 I vs Placebo; Test type: Superiority; p = 0.0987, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: SUNPG1623 II vs Placebo; Test type: Superiority; p = 0.0360, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: SUNPG1623 Dose III vs Placebo; Test type: Superiority; p = 0.0346, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: SUNPG1623 Dose IV vs Placebo; Test type: Superiority; p = 0.4442, Cochran-Mantel-Haenszel

16. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire- Disability Index
Description: as for outcome 15
Time Frame: Week 52
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score for the disability index
Groups:
- SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24: Group: SUNPG1623 IV dosage: Mid to long-term dose dosage form: subcutaneous injection frequency of administration: q12 weeks.
  Subjects who received SUNPG1623 Dose IV during Part 1 but failed to show clinical response to treatment at Week 24 entered Part 2 and received SUNPG1623 II until Week 48
Arm/Group | SUNPG1623 I | SUNPG1623 II | SUNPG1623 Dose III | SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24 | Placebo Moved to SUNPG1623 II After Week 24
Number analyzed (Participants) | 78 | 79 | 77 | 78 | 79
score for the disability index | -0.4869 (0.52093) | -0.5430 (0.59145) | -0.4857 (0.56968) | -0.4583 (0.52285) | -0.4700 (0.54013)
Statistical Analysis 1: Comparison: SUNPG1623 I; Test type: Superiority; Mean Difference (Net) = -0.4869, Standard Deviation 0.52093
Statistical Analysis 2: Comparison: SUNPG1623 II; Test type: Superiority; Mean Difference (Net) = -0.5430, Standard Deviation 0.59145
Statistical Analysis 3: Comparison: SUNPG1623 Dose III; Test type: Superiority; Mean Difference (Net) = -0.4857, Standard Deviation 0.56968
Statistical Analysis 4: Comparison: SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24; Test type: Superiority; Mean Difference (Net) = -0.4583, Standard Deviation 0.52285
Statistical Analysis 5: Comparison: Placebo Moved to SUNPG1623 II After Week 24; Test type: Superiority; Mean Difference (Net) = -0.4700, Standard Deviation 0.54013

17. Secondary Outcome: Acute Phase C - Reactive Protein
Description: C-reactive protein (CRP) is a blood test marker for inflammation in the body. CRP is produced in the liver and its level is measured by testing the blood.
  CRP is classified as an acute phase reactant, which means that its levels will rise in response to inflammation
Time Frame: week 1, week 4, week 8, week 12, week 16, week 20, and week 24
Population: Statistical Analysis (Mixed Model Repeated Measures) of Change From Baseline in CRP (mg/L) up to Week 24 - (No Imputation) Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | SUNPG1623 I | SUNPG1623 II | SUNPG1623 Dose III | SUNPG1623 Dose IV | Placebo
Number analyzed (Participants) | 77 | 78 | 76 | 78 | 79
mg/L
  Week 1 | 0.19 (0.967) | -0.75 (0.961) | -0.50 (0.979) | 2.08 (0.961) | 0.51 (0.964)
  Week 4 | -0.71 (1.239) | -3.41 (1.227) | -0.82 (1.223) | 0.64 (1.222) | -0.28 (1.206)
  Week 8 | -2.96 (1.506) | -3.21 (1.476) | -1.54 (1.502) | 1.95 (1.495) | 1.24 (1.465)
  Week 12 | -2.21 (1.121) | -3.04 (1.097) | -2.59 (1.104) | 0.11 (1.124) | 1.49 (1.097)
  Week 16 | -3.37 (1.505) | -3.57 (1.462) | -1.67 (1.485) | -1.58 (1.505) | 2.25 (1.474)
  Week 20 | -3.72 (1.708) | -2.76 (1.656) | -2.57 (1.677) | -0.61 (1.715) | 4.60 (1.672)
  Week 24 | -3.56 (1.088) | -2.33 (1.054) | -3.23 (1.071) | -2.06 (1.088) | 0.55 (1.065)
Statistical Analysis 1: Comparison: SUNPG1623 I vs Placebo; Test type: Superiority; p = 0.0064, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: SUNPG1623 II vs Placebo; Test type: Superiority; p = 0.0516, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: SUNPG1623 Dose III vs Placebo; Test type: Superiority; p = 0.0114, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: SUNPG1623 Dose IV vs Placebo; Test type: Superiority; p = 0.0820, Cochran-Mantel-Haenszel

18. Secondary Outcome: Acute Phase C - Reactive Protein
Description: C-reactive protein (CRP) is a blood test marker for inflammation in the body. CRP is produced in the liver and its level is measured by testing the blood.
  CRP is classified as an acute phase reactant, which means that its levels will rise in response to inflammation.
  Change from Baseline in C-Reactive Protein.
Time Frame: Week 52
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | SUNPG1623 I | SUNPG1623 II | SUNPG1623 Dose III | SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24 | Placebo Moved to SUNPG1623 II After Week 24
Number analyzed (Participants) | 78 | 79 | 77 | 78 | 79
mg/L | -3.43 (12.506) | -3.68 (10.770) | -6.05 (19.004) | -4.61 (9.508) | -6.75 (19.649)
Statistical Analysis 1: Comparison: SUNPG1623 I; Test type: Superiority; Mean Difference (Net) = -3.43, Standard Deviation 12.506
Statistical Analysis 2: Comparison: SUNPG1623 II; Test type: Superiority; Mean Difference (Net) = -3.68, Standard Deviation 10.770
Statistical Analysis 3: Comparison: SUNPG1623 Dose III; Test type: Superiority; Mean Difference (Net) = -6.05, Standard Deviation 19.004
Statistical Analysis 4: Comparison: SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24; Test type: Superiority; Mean Difference (Net) = -4.61, Standard Deviation 9.508
Statistical Analysis 5: Comparison: Placebo Moved to SUNPG1623 II After Week 24; Test type: Superiority; Mean Difference (Net) = -6.75, Standard Deviation 19.649

19. Secondary Outcome: Erythrocyte Sedimentation Rate
Description: An erythrocyte sedimentation rate (ESR) is a type of blood test that measures how quickly erythrocytes (red blood cells) settle at the bottom of a test tube that contains a blood sample. This test help determine if you have a condition that causes inflammation.
Time Frame: week 1, week 4, week 8, week 12, week 16, week 20, and week 24
Population: Statistical Analysis (Mixed Model Repeated Measures) of Change From Baseline in ESR (mm/hr) up to Week 24 - (No Imputation) Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: mm/hr
Arm/Group | SUNPG1623 I | SUNPG1623 II | SUNPG1623 Dose III | SUNPG1623 Dose IV | Placebo
Number analyzed (Participants) | 70 | 68 | 69 | 68 | 62
mm/hr
  Week 1 | -3.1 (1.39) | -3.0 (1.40) | -3.3 (1.41) | -1.1 (1.41) | -2.6 (1.45)
  Week 4 | -6.9 (1.46) | -5.9 (1.48) | -5.5 (1.45) | -5.6 (1.47) | -4.8 (1.51)
  Week 8 | -8.7 (1.58) | -6.5 (1.58) | -7.1 (1.58) | -5.5 (1.60) | -3.6 (1.64)
  Week 12 | -8.6 (1.59) | -6.8 (1.59) | -7.9 (1.58) | -6.6 (1.62) | -2.3 (1.66)
  Week 16 | -9.4 (1.93) | -8.4 (1.92) | -8.3 (1.91) | -6.0 (1.96) | -3.3 (2.02)
  Week 20 | -9.6 (1.73) | -7.2 (1.72) | -9.2 (1.71) | -8.5 (1.76) | -4.4 (1.81)
  Week 24 | -8.0 (1.86) | -6.9 (1.85) | -8.2 (1.84) | -8.7 (1.89) | -2.3 (1.95)
Statistical Analysis 1: Comparison: SUNPG1623 I vs Placebo; Test type: Superiority; p = 0.0351, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: SUNPG1623 II vs Placebo; Test type: Superiority; p = 0.0876, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: SUNPG1623 Dose III vs Placebo; Test type: Superiority; p = 0.0269, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: SUNPG1623 Dose IV vs Placebo; Test type: Superiority; p = 0.0185, Cochran-Mantel-Haenszel

20. Secondary Outcome: Change From Baseline in Erythrocyte Sedimentation Rate
Description: as for outcome 19
Time Frame: Week 52
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | SUNPG1623 I | SUNPG1623 II | SUNPG1623 Dose III | SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24 | Placebo Moved to SUNPG1623 II After Week 24
Number analyzed (Participants) | 78 | 79 | 77 | 78 | 79
mm/hr | -7.2 (19.58) | -7.2 (15.26) | -8.9 (20.48) | -9.7 (19.02) | -9.2 (20.47)
Statistical Analysis 1: Comparison: SUNPG1623 I; Test type: Superiority; Mean Difference (Net) = -7.2, Standard Deviation 19.58
Statistical Analysis 2: Comparison: SUNPG1623 II; Test type: Superiority; Mean Difference (Net) = -7.2, Standard Deviation 15.26
Statistical Analysis 3: Comparison: SUNPG1623 Dose III; Test type: Superiority; Median Difference (Net) = -8.9, Standard Deviation 20.48
Statistical Analysis 4: Comparison: SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24; Test type: Superiority; Mean Difference (Net) = -9.7, Standard Deviation 19.02
Statistical Analysis 5: Comparison: Placebo Moved to SUNPG1623 II After Week 24; Test type: Superiority; Mean Difference (Net) = -9.2, Standard Deviation 20.47

21. Secondary Outcome: The Proportion of Subjects Who Require Adjustment of Background Therapy
Time Frame: Week 16
Population: Subjects Who Require Adjustment of Background Therapy at Week 16 Full Analysis Set
Measure: Number; unit: proportion of subjects
Arm/Group | SUNPG1623 I | SUNPG1623 II | SUNPG1623 Dose III | SUNPG1623 Dose IV | Placebo
Number analyzed (Participants) | 78 | 79 | 77 | 78 | 79
proportion of subjects | 0 | 0.0127 | 0.0130 | 0.0256 | 0.0127
Statistical Analysis 1: Comparison: SUNPG1623 I vs Placebo; Test type: Superiority; Proportion with Adjustment of Background = 1.27, 95% CI 2-sided [0.00 to 3.73], Standard Error of Mean 1.26
Statistical Analysis 2: Comparison: SUNPG1623 II vs Placebo; Test type: Superiority; Proportion with Adjustment of Background = 1.30, 95% CI 2-sided [0.00 to 3.83], Standard Error of Mean 1.29
Statistical Analysis 3: Comparison: SUNPG1623 Dose III vs Placebo; Test type: Superiority; Proportion with Adjustment of Background = 2.56, 95% CI 2-sided [0.00 to 6.07], Standard Error of Mean 1.79
Statistical Analysis 4: Comparison: SUNPG1623 Dose IV vs Placebo; Test type: Superiority; Proportion with Adjustment of Background = 1.27, 95% CI 2-sided [0.00 to 3.73], Standard Error of Mean 1.26

22. Secondary Outcome: Disease Activity Score (DAS) 28 (Joints) C - Reactive Protein (DAS28-CRP) Response Rate
Description: The Disease Activity Score 28-item C-Reactive Protein: assessed across 28 joints including the shoulder, elbow, wrist, MCP (1 through 5), PIP (1 through 5) and knee, with all 14 joints assessed for each side of the body. It is a composite score derived from examination of the 28 joints for swelling and tenderness, global assessment of pain and overall status using a VAS and a blood marker of inflammation (hsCRP).
  DAS28-CRP(4) = 0.56*sqrt(TJC28) + 0.28*sqrt(SJC28) + 0.36*ln(CRP+1) + 0.014*GH + 0.96 TJC- tender joint count, SJC- swollen joint count, CRP- C reactive protein, GH - patient global health
Time Frame: week 1, week 4, week 8, week 12, week 16, week 20, week 24 and Week 52
Population: Cochran-Mantel-Haenszel Analysis of DAS28-CRP Response Rates up to Week 24 Full Analysis Set.
  DAS28-CRP Response Rates up to Week 52-Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SUNPG1623 I | SUNPG1623 II | SUNPG1623 Dose III | SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24 | Placebo Moved to SUNPG1623 II After Week 24
Number analyzed (Participants) | 78 | 79 | 77 | 78 | 79
percentage of participants
  Week 1 | 11.54 | 12.66 | 10.39 | 5.13 | 6.33
  Week 4 | 20.51 | 17.72 | 15.58 | 15.38 | 13.92
  Week 8 | 35.90 | 29.11 | 29.87 | 23.08 | 18.99
  Week 12 | 38.46 | 40.51 | 31.17 | 29.49 | 18.99
  Week 16 | 48.72 | 48.10 | 36.36 | 35.90 | 13.92
  Week 20 | 60.26 | 60.76 | 37.66 | 43.59 | 21.52
  Week 24 | 58.97 | 64.56 | 58.44 | 53.85 | 30.38
  Week 52: number analyzed (Participants) | 67 | 64 | 59 | 76 | 75
  Week 52 | 85.07 | 81.25 | 76.27 | 71.05 | 65.33
Statistical Analysis 1: Comparison: SUNPG1623 I; Test type: Superiority; % response rate = 85.07, 95% CI 2-sided [76.54 to 93.61], Standard Error of Mean 4.35
Statistical Analysis 2: Comparison: SUNPG1623 II; Test type: Superiority; % response rate = 81.25, 95% CI 2-sided [71.69 to 90.81], Standard Error of Mean 4.88
Statistical Analysis 3: Comparison: SUNPG1623 Dose III; Test type: Superiority; % response rate = 76.27, 95% CI 2-sided [65.42 to 87.13], Standard Error of Mean 5.54
Statistical Analysis 4: Comparison: SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24; Test type: Superiority; % response rate = 71.05, 95% CI 2-sided [60.86 to 81.25], Standard Error of Mean 5.20
Statistical Analysis 5: Comparison: Placebo Moved to SUNPG1623 II After Week 24; Test type: Superiority; % response rate = 65.33, 95% CI 2-sided [54.56 to 76.10], Standard Error of Mean 5.50

23. Secondary Outcome: Minimal Disease Activity
Description: A psoriatic arthritis patient is defined as having a Minimal Disease Activity (MDA) response (Yes/No) when the patient meets at least 5 of the 7 following criteria:
  1. tender joint count ≤1;
  2. swollen joint count ≤1;
  3. PASI score ≤1 or BSA ≤3%;
  4. patient Arthritis Pain (VAS)
     ≤15 mm;
  5. patient's global arthritis assessment (VAS) ≤20 mm;
  6. HAQ-DI score ≤0.5;
  7. tender entheseal points (using LEI) ≤1.
Time Frame: week 1, week 4, week 8, week 12, week 16, week 20, week 24 and week 52
Population: Cochran-Mantel-Haenszel Analysis of MDA Response Rates up to Week 24 (Missing Response = Non-response) Full Analysis Set.
  MDA Response Rates up to Week 52- Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SUNPG1623 I | SUNPG1623 II | SUNPG1623 Dose III | SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24 | Placebo Moved to SUNPG1623 II After Week 24
Number analyzed (Participants) | 78 | 79 | 77 | 78 | 79
percentage of participants
  Week 1 | 0 | 1.27 | 0 | 0 | 0
  Week 4 | 3.85 | 1.27 | 1.30 | 2.56 | 1.27
  Week 8 | 3.85 | 2.53 | 2.60 | 0 | 2.53
  Week 12 | 12.82 | 8.86 | 7.79 | 8.97 | 2.53
  Week 16 | 12.82 | 6.33 | 7.79 | 8.97 | 1.27
  Week 20 | 17.95 | 15.19 | 9.09 | 8.97 | 2.53
  Week 24 | 33.33 | 34.18 | 28.57 | 19.23 | 6.33
  week 52: number analyzed (Participants) | 65 | 59 | 60 | 68 | 69
  week 52 | 56.92 | 64.41 | 45.00 | 47.06 | 42.03
Statistical Analysis 1: Comparison: SUNPG1623 I; Test type: Superiority; % response rate = 56.92, 95% CI 2-sided [44.88 to 68.96], Standard Error of Mean 6.14
Statistical Analysis 2: Comparison: SUNPG1623 II; Test type: Superiority; % response rate = 64.41, 95% CI 2-sided [52.19 to 76.62], Standard Error of Mean 6.23
Statistical Analysis 3: Comparison: SUNPG1623 Dose III; Test type: Superiority; % response rate = 45.00, 95% CI 2-sided [32.41 to 57.59], Standard Error of Mean 6.42
Statistical Analysis 4: Comparison: SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24; Test type: Superiority; % response rate = 47.06, 95% CI 2-sided [35.20 to 58.92], Standard Error of Mean 6.05
Statistical Analysis 5: Comparison: Placebo Moved to SUNPG1623 II After Week 24; Test type: Superiority; % response rate = 42.03, 95% CI 2-sided [30.38 to 53.68], Standard Error of Mean 5.94

24. Secondary Outcome: Change From Baseline in Leeds Dactylitis Index (LDI)
Description: tenderness score (0 = no tenderness, 1 = tender, 2 = tender and wince, and 3 = tender and withdraw)
  Total score= {[Circumference involved digit/ Circumference contralateral Digit (or Tables)] - 1x 100}x Tenderness score
  Standard reference: Hands Digit Men Women Thumb 70 58 Index 63 54 Middle 63 54 Ring 59 50 Little 52 44 Standard reference: Feet Digit Men Women Great Toe 82 72 Second 52 46 Middle 50 44 Fourth 50 44 Little 52 45
  The difference between circumference of affected finger and contralateral not affected digit cannot be defined for maximum value. Therefore, it is difficult to provide scale range for the final score. No theoretical range exists for the Leeds Dactylitis Index.
  Lower Leeds Dactylitis Index score represent better outcome.
Time Frame: week 4, week 12, and week 24
Population: Statistical Analysis (Mixed Model Repeated Measures) of Change From Baseline in LDI up to Week 24 - (No Imputation) Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | SUNPG1623 I | SUNPG1623 II | SUNPG1623 Dose III | SUNPG1623 Dose IV | Placebo
Number analyzed (Participants) | 53 | 56 | 46 | 48 | 54
score on a scale
  Week 4 | -17.385 (9.8336) | -17.918 (9.5818) | -19.150 (10.4630) | -5.385 (10.2843) | 19.891 (9.6640)
  Week 12 | -21.041 (7.8359) | -23.163 (7.5635) | -23.948 (8.3579) | -9.982 (8.2513) | -2.990 (7.7362)
  Week 24 | -22.987 (3.5112) | -25.123 (3.2307) | -27.572 (3.5088) | -19.873 (3.4520) | -24.706 (3.2252)
Statistical Analysis 1: Comparison: SUNPG1623 I vs Placebo; Test type: Superiority; p = 0.7081, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: SUNPG1623 II vs Placebo; Test type: Superiority; p = 0.9244, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: SUNPG1623 Dose III vs Placebo; Test type: Superiority; p = 0.5365, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: SUNPG1623 Dose IV vs Placebo; Test type: Superiority; p = 0.2925, Cochran-Mantel-Haenszel

25. Secondary Outcome: Change From Baseline in Leeds Dactylitis Index (LDI)
Description: as for outcome 24
Time Frame: Week 52
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SUNPG1623 I | SUNPG1623 II | SUNPG1623 Dose III | SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24 | Placebo Moved to SUNPG1623 II After Week 24
Number analyzed (Participants) | 78 | 79 | 77 | 78 | 79
score on a scale | -14.453 (31.9358) | -18.883 (57.1147) | -27.084 (76.2272) | -26.173 (87.5367) | -50.399 (141.6770)
Statistical Analysis 1: Comparison: SUNPG1623 I; Test type: Superiority; Mean Difference (Net) = -14.453, Standard Deviation 31.9358
Statistical Analysis 2: Comparison: SUNPG1623 II; Test type: Superiority; Mean Difference (Net) = -18.883, Standard Deviation 57.1147
Statistical Analysis 3: Comparison: SUNPG1623 Dose III; Test type: Superiority; Mean Difference (Net) = -27.084, Standard Deviation 76.2272
Statistical Analysis 4: Comparison: SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24; Test type: Superiority; Mean Difference (Net) = -26.173, Standard Deviation 87.5367
Statistical Analysis 5: Comparison: Placebo Moved to SUNPG1623 II After Week 24; Test type: Superiority; Mean Difference (Net) = -50.399, Standard Deviation 141.6770

26. Secondary Outcome: Change From Baseline in Leeds Enthesitis Index (LEI)
Description: The LEI examines tenderness at 6 sites:
  2 sites (left and right) at each of the lateral epicondyles of the humerus, medial condyles of the femur and the insertion of the Achilles tendon. For each entheseal site, assessment is made of the adjacent joint in terms of tenderness and soft-tissue swelling, with a score of 1 if present. The LEI score range is 0-6.
  Lower the score better is the outcome
Time Frame: week 4, week 12 and week 24
Population: Statistical Analysis (Mixed Model Repeated Measures) of Change From Baseline in LEI up to Week 24 - (No Imputation) Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | SUNPG1623 I | SUNPG1623 II | SUNPG1623 Dose III | SUNPG1623 Dose IV | Placebo
Number analyzed (Participants) | 72 | 77 | 75 | 76 | 78
score on a scale
  Week 4 | -0.5 (0.15) | -0.4 (0.14) | -0.5 (0.14) | -0.4 (0.14) | -0.4 (0.14)
  Week 12 | -0.8 (0.15) | -0.7 (0.14) | -0.9 (0.15) | -0.8 (0.15) | -0.7 (0.14)
  Week 24 | -1.3 (0.16) | -0.9 (0.15) | -1.2 (0.15) | -1.1 (0.15) | -0.8 (0.15)
Statistical Analysis 1: Comparison: SUNPG1623 I vs Placebo; Test type: Superiority; p = 0.0203, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: SUNPG1623 II vs Placebo; Test type: Superiority; p = 0.5194, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: SUNPG1623 Dose III vs Placebo; Test type: Superiority; p = 0.0599, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: SUNPG1623 Dose IV vs Placebo; Test type: Superiority; p = 0.1220, Cochran-Mantel-Haenszel

27. Secondary Outcome: Change From Baseline in Leeds Enthesitis Index (LEI)
Description: as for outcome 26
Time Frame: Week 52
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SUNPG1623 I | SUNPG1623 II | SUNPG1623 Dose III | SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24 | Placebo Moved to SUNPG1623 II After Week 24
Number analyzed (Participants) | 78 | 79 | 77 | 78 | 79
score on a scale | -1.3 (1.86) | -1.0 (1.56) | -1.7 (2.08) | -1.2 (1.75) | -1.2 (1.82)
Statistical Analysis 1: Comparison: SUNPG1623 I; Test type: Superiority; Mean Difference (Net) = -1.3, Standard Deviation 1.86
Statistical Analysis 2: Comparison: SUNPG1623 II; Test type: Superiority; Mean Difference (Net) = -1.0, Standard Deviation 1.56
Statistical Analysis 3: Comparison: SUNPG1623 Dose III; Test type: Superiority; Mean Difference (Net) = -1.7, Standard Deviation 2.08
Statistical Analysis 4: Comparison: SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24; Test type: Superiority; Mean Difference (Net) = -1.2, Standard Deviation 1.75
Statistical Analysis 5: Comparison: Placebo Moved to SUNPG1623 II After Week 24; Test type: Superiority; Mean Difference (Net) = -1.2, Standard Deviation 1.82

ADVERSE EVENTS:
Time Frame: 72 week
Groups:
- Part 1: SUNPG1623 I; Part 2: SUNPG1623 I: Group: SUNPG1623 I dosage: Short-term dose dosage form: subcutaneous injection frequency of administration: q4 weeks
- Part 1 : SUNPG1623 II; Part 2 : SUNPG1623 II: Group: SUNPG1623 II dosage: Mid-term dose dosage form: subcutaneous injection frequency of administration: q12 weeks
- Part 1 : SUNPG1623 Dose III; Part 2 : SUNPG1623 Dose III: Group: SUNPG1623 III dosage: Mid-term dose dosage form: subcutaneous injection frequency of administration: q12 weeks
- Part 1 : SUNPG1623 Dose IV: Group: SUNPG1623 IV dosage: Mid to long-term dose dosage form: subcutaneous injection frequency of administration: q12 weeks
  Subjects who received SUNPG1623 Dose IV during Part 1 but failed to show clinical response to treatment at Week 24 entered Part 2 and received SUNPG1623 II until Week 48
- Part 1 : Placebo: Group: Placebo dosage: Mid to long-term dose dosage form: subcutaneous injection frequency of administration: q12 weeks
  Subjects who received placebo during Part 1 but failed to show clinical response to treatment at Week 24 entered Part 2 and received SUNPG1623 II until Week 48
- Part 2: Week 24 - 48: SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24: Subjects who received SUNPG1623 Dose IV during Part 1 but failed to show clinical response to treatment at Week 24 entered Part 2 and received SUNPG1623 II until Week 48
- Part 2: Week 24 - 48: Placebo Moved to SUNPG1623 II After Week 24: Subjects who received placebo during Part 1 but failed to show clinical response to treatment at Week 24 entered Part 2 and received SUNPG1623 II until Week 48
- Part 3: SUNPG1623 I; Part 3 : SUNPG1623 II; Part 3 : SUNPG1623 Dose III: Wash-out period
- Part 3 :Wash-out Period (SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24): Group: SUNPG1623 IV dosage: Mid to long-term dose dosage form: subcutaneous injection frequency of administration: q12 weeks
  Part 2 : Subjects who received SUNPG1623 Dose IV during Part 1 but failed to show clinical response to treatment at Week 24 entered Part 2 and received SUNPG1623 II until Week 48
  Part 3 : wash-out period
- Part 3 : Wash-out Period (Placebo Moved to SUNPG1623 II After Week 24): Group: Placebo dosage: Mid to long-term dose dosage form: subcutaneous injection frequency of administration: q12 weeks
  Part 2 : Subjects who received placebo during Part 1 but failed to show clinical response to treatment at Week 24 entered Part 2 and received SUNPG1623 II until Week 48
  Part 3 : wash-out period
Arm/Group | Part 1: SUNPG1623 I | Part 1 : SUNPG1623 II | Part 1 : SUNPG1623 Dose III | Part 1 : SUNPG1623 Dose IV | Part 1 : Placebo | Part 2: SUNPG1623 I | Part 2 : SUNPG1623 II | Part 2 : SUNPG1623 Dose III | Part 2: Week 24 - 48: SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24 | Part 2: Week 24 - 48: Placebo Moved to SUNPG1623 II After Week 24 | Part 3: SUNPG1623 I | Part 3 : SUNPG1623 II | Part 3 : SUNPG1623 Dose III | Part 3 :Wash-out Period (SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24) | Part 3 : Wash-out Period (Placebo Moved to SUNPG1623 II After Week 24)
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/79 | 0/77 | 0/78 | 0/79 | 0/78 | 0/79 | 0/77 | 0/78 | 0/79 | 1/78 | 0/79 | 0/77 | 0/78 | 0/79
Serious Adverse Events (participants affected / at risk) | 2/78 | 2/79 | 2/77 | 1/78 | 2/79 | 0/78 | 0/79 | 0/77 | 3/78 | 1/79 | 3/78 | 1/79 | 1/77 | 1/78 | 2/79
Other Adverse Events (participants affected / at risk) | 17/78 | 18/79 | 16/77 | 22/78 | 18/79 | 14/78 | 11/79 | 6/77 | 18/78 | 9/79 | 8/78 | 1/79 | 3/77 | 8/78 | 8/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: SUNPG1623 I (N=78) | Part 1 : SUNPG1623 II (N=79) | Part 1 : SUNPG1623 Dose III (N=77) | Part 1 : SUNPG1623 Dose IV (N=78) | Part 1 : Placebo (N=79) | Part 2: SUNPG1623 I (N=78) | Part 2 : SUNPG1623 II (N=79) | Part 2 : SUNPG1623 Dose III (N=77) | Part 2: Week 24 - 48: SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24 (N=78) | Part 2: Week 24 - 48: Placebo Moved to SUNPG1623 II After Week 24 (N=79) | Part 3: SUNPG1623 I (N=78) | Part 3 : SUNPG1623 II (N=79) | Part 3 : SUNPG1623 Dose III (N=77) | Part 3 :Wash-out Period (SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24) (N=78) | Part 3 : Wash-out Period (Placebo Moved to SUNPG1623 II After Week 24) (N=79)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst ruptured (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toxicity to various agents (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple sclerosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: SUNPG1623 I (N=78) | Part 1 : SUNPG1623 II (N=79) | Part 1 : SUNPG1623 Dose III (N=77) | Part 1 : SUNPG1623 Dose IV (N=78) | Part 1 : Placebo (N=79) | Part 2: SUNPG1623 I (N=78) | Part 2 : SUNPG1623 II (N=79) | Part 2 : SUNPG1623 Dose III (N=77) | Part 2: Week 24 - 48: SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24 (N=78) | Part 2: Week 24 - 48: Placebo Moved to SUNPG1623 II After Week 24 (N=79) | Part 3: SUNPG1623 I (N=78) | Part 3 : SUNPG1623 II (N=79) | Part 3 : SUNPG1623 Dose III (N=77) | Part 3 :Wash-out Period (SUNPG1623 Dose IV Moved to SUNPG1623 II After Week 24) (N=78) | Part 3 : Wash-out Period (Placebo Moved to SUNPG1623 II After Week 24) (N=79)
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 7 | 1 | 4 | 5 | 5 | 2 | 2 | 2 | 7 | 3 | 2 | 0 | 1 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 4 | 3 | 3 | 1 | 3 | 4 | 2 | 4 | 0 | 0 | 0 | 1 | 2 | 0
Headache (Nervous system disorders) | 4 | 1 | 5 | 5 | 3 | 1 | 3 | 2 | 0 | 1 | 3 | 0 | 1 | 1 | 2
Sleep Disorder (Psychiatric disorders) | 1 | 5 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 3 | 6 | 1 | 2 | 5 | 4 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 3 | 1 | 3 | 1 | 1 | 0 | 4 | 1 | 0 | 0 | 0 | 3 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 4 | 2 | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-03-16): https://cdn.clinicaltrials.gov/large-docs/92/NCT02980692/Prot_002.pdf
  • Statistical Analysis Plan (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/92/NCT02980692/SAP_003.pdf